CLINICAL TRIAL: NCT00525590
Title: A Phase 2, Multicenter, Exploratory Study, Evaluating the Treatment Effect of Surgery Plus GLIADEL® Wafer in Patients With Metastatic Brain Cancer
Brief Title: Exploratory Study, Evaluating the Treatment Effect of Surgery Plus GLIADEL® Wafer in Patients With Metastatic Brain Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GLIA-001
Record Dates: First submitted 2007-09-04; First posted 2007-09-06 (Estimated); Results first posted 2020-03-16 (Actual); Last update posted 2020-03-16 (Actual); Status verified 2020-02

CONDITIONS: Metastatic Brain Cancer
Keywords: Gliadel
MeSH Terms: conditions — Brain Neoplasms | interventions — carmustine, poliferprosan 20 drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: GLIADEL

INTERVENTIONS:
Drug: GLIADEL — Resect the tumor as completely as possible. After repeated irrigation of the decompressed area demonstrates no bleeding, and care is taken not to have any foreign material enter the ventricle, up to 8 GLIADEL wafers should be placed to cover the entire surface area of the resection cavity (if possible). Slight overlapping of wafer edges is permitted. The number of wafers will be determined by the size of the tumor resection cavity. Each GLIADEL wafer contains 7.7 mg of carmustine, resulting in a dose of 61.6 mg when 8 wafers are implanted. The GLIADEL wafer is a round white to yellow disk with flat surfaces.

SUMMARY:
The purpose of this study is to determine the effect of the surgical intervention and insertion of GLIADEL wafers on the neurocognitive functioning in patients with metastatic brain cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Can provide signed/dated Informed Consent, and Health Insurance Portability and Accountability Act of 1996 (HIPAA) authorization.
2. Are a male or female patient 18 years of age or older.
3. Are willing to a use barrier method of contraception if fertile or of childbearing potential until 30 days after surgical resection. If the patient receives subsequent chemotherapy during study participation (as allowed by the protocol), appropriate contraception will be managed by the principal investigator.
4. Have a primary diagnosis of solid-based tumor cancer (except small cell lung cancer (SCLS), lymphoma, germ cell cancer or anaplastic thyroid cancer) or unknown primary cancer and have 1-3 brain metastasis(es) for which surgical resection is planned for a single metastasis and any remaining metastases are planned for stereotactic radiosurgery (SRS);

   OR

   an intra-operative diagnosis of metastatic brain tumor in a patient with a single brain lesion.
5. Have a life expectancy of ≥12 weeks.
6. Have a Karnofsky Performance Status (KPS) score of 70 or higher.
7. Have Recursive Partitioning Analysis (RPA) status of 1 or 2.
8. Women of childbearing potential must have a negative serum or urine pregnancy test within 14 days of the surgical resection; and
9. Patients must be able to understand English, either orally or in writing, and be able to consent and complete the required assessments and procedures.

Exclusion Criteria:

1. Are unable or unwilling to understand study assessment or to cooperate with the study procedures as determined by the investigator.
2. Have a history of allergic reaction or known hypersensitivity to BCNU (carmustine) or other components of the GLIADEL, such as polifeprosan polymer.
3. Have a history of prior cranial irradiation.
4. Have a prior diagnosis of Central Nervous System (CNS) tumor.
5. Have received prior treatment for brain tumors.
6. Have had prior exposure to GLIADEL or its components, such as polifeprosan polymer.
7. Have any uncontrolled medical or psychiatric conditions which preclude them from participating in or completing the study procedures.
8. Concurrent severe medical conditions include, but are not limited to, active infection, acute hepatitis, cardiac arrhythmia, unstable angina, congestive heart failure, uncontrolled diabetes mellitus, uncontrolled seizures, pulmonary insufficiency, pulmonary fibrosis, pulmonary embolus, etc.
9. Have a diagnosis of tumor in the brain stem or posterior fossa.
10. Have an RPA status of 3.
11. Have a diagnosis of leptomeningeal disease at time of enrollment; or
12. Are currently pregnant or lactating, or plan to become pregnant during the course of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2007-12-12 (Actual); Primary Completion 2010-12-01 (Actual); Study Completion 2010-12-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (17):
- United States (17):
  - University of Arizona / University Medical Center, Tucson, Arizona
  - University of California, Los Angeles, Los Angeles, California
  - University of South Florida, Tampa, Florida
  - H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida
  - The University of Chicago, Chicago, Illinois
  - NorthShore University HealthSystem Reseach Institute, Evanston, Illinois
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Weill Medical College Department of Neurological Surgery, New York, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Carolina Neurosurgery & Spine Associates, Charlotte, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - The Ohio State University Medical Center, Columbus, Ohio
  - Temple University, Philadelphia, Pennsylvania
  - Methodist University Hospital, Memphis, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - UT Southwestern Medical Center at Dallas, Dallas, Texas
  - Trinity Mother Frances Health System, Tyler, Texas

REFERENCES:
- [Derived] Brem S, Meyers CA, Palmer G, Booth-Jones M, Jain S, Ewend MG. Preservation of neurocognitive function and local control of 1 to 3 brain metastases treated with surgery and carmustine wafers. Cancer. 2013 Nov 1;119(21):3830-8. doi: 10.1002/cncr.28307. Epub 2013 Aug 23. PMID 24037801

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 12 sites in the United States from 12 December 2007 to 01 December 2010.
Pre-assignment Details: A total of 82 participants with metastatic brain cancer were screened, of which 69 participants were enrolled and 59 participants were treated.
Groups:
- GLIADEL: Participants with metastatic brain tumors who underwent neurosurgical resection of their lesions were implanted with up to 8 GLIADEL wafers in their tumor cavities (each containing 7.7 [milligram] mg of carmustine). Participants were followed up to 12 months or until the participant experienced local recurrence, withdrew, died, was lost to follow-up, or the study was closed.
Period: Overall Study
Arm/Group | GLIADEL
Started | 59
Completed | 14
Not Completed | 45
Not completed — Adverse Event | 3
Not completed — Physician Decision | 3
Not completed — Withdrawal by Subject | 16
Not completed — Lost to Follow-up | 1
Not completed — Death | 9
Not completed — Other | 13

BASELINE CHARACTERISTICS:
Population: The safety analysis set included all enrolled participants who underwent surgical resection and received GLIADEL treatment.
Groups:
- GLIADEL: Participants with metastatic brain tumors who underwent neurosurgical resection of their lesions were implanted with up to 8 GLIADEL wafers in their tumor cavities (each containing 7.7 mg of carmustine). Participants were followed up to 12 months or until the participant experienced local recurrence, withdrew, died, was lost to follow-up, or the study was closed.
Arm/Group | GLIADEL
Number analyzed (Participants) | 59
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.0 (11.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33
  Male | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 59
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 55
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Rate of Deterioration in Neurocognitive Functioning (NF) at Month 12
Description: NF was assessed as the performance of 3 neurocognitive domains:memory(MD),executive function(EFD), fine motor coordination(FMCD). For each domain, z-scores were derived from participant's scores in individual neurocognitive tests using an age-adjusted and education-adjusted normative distribution of scores from an unimpaired population.Individual z-scores from related tests were averaged to determine overall z-score.If a z-score average decreased from baseline by greater than or equal to(>=)3 standard deviations(SD)in tests' normative age-adjusted distribution on 2 consecutive visits or decreased by >=3 SD on last follow-up visit, participant were considered to have significant deterioration in their NF at time of the first decrease in z-score.Deterioration in NF:demonstrated deterioration for at least two of the three neurocognitive domains based on these changes from screening.Rate of deterioration in NF was measured as estimated percentage of participants using Kaplan-Meier method.
Time Frame: Month 12
Population: The per protocol 1 (PP1) population included all participants who received surgery plus GLIADEL, had an intra-operative diagnosis confirmed by permanent pathology findings, remained compliant with protocol procedures, and did not receive disallowed concomitant therapies (example whole brain radiation therapy [WBRT]) before recurrence.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- GLIADEL: Participants with metastatic brain tumors who underwent neurosurgical resection of their lesions were implanted with up to 8 GLIADEL wafers in their tumor cavities (each containing 7.7 mg of carmustine).
Arm/Group | GLIADEL
Number analyzed (Participants) | 54
percentage of participants | 2.8 [0.40 to 18.13]

2. Primary Outcome: Number of Participants With Neurocognitive Domains Preserved at Month 2
Description: Preservation of NF was defined as a decrease of <=1 SD, any increase, or no change (0 SD) in z-score for each domain (memory domain, executive function domain, and fine motor coordination domain).
Time Frame: Month 2
Population: The PP1 population included all participants who received surgery plus GLIADEL, had an intra-operative diagnosis confirmed by permanent pathology findings, remained compliant with protocol procedures, and did not receive disallowed concomitant therapies (example WBRT) before recurrence.
Measure: Count of Participants; unit: Participants
Arm/Group | GLIADEL
Number analyzed (Participants) | 54
Participants
  Domains preserved=3 | 26
  Domains preserved=2 | 12
  Domains preserved=1 | 4
  Domains preserved=0 | 3

3. Primary Outcome: Number of Participants With Neurocognitive Domains Preserved at Month 4
Description: as for outcome 2
Time Frame: Month 4
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | GLIADEL
Number analyzed (Participants) | 54
Participants
  Domains preserved=3 | 24
  Domains preserved=2 | 9
  Domains preserved=1 | 2
  Domains preserved=0 | 1

4. Primary Outcome: Number of Participants With Neurocognitive Domains Preserved at Month 6
Description: as for outcome 2
Time Frame: Month 6
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | GLIADEL
Number analyzed (Participants) | 54
Participants
  Domains preserved=3 | 17
  Domains preserved=2 | 5
  Domains preserved=1 | 2
  Domains preserved=0 | 0

5. Primary Outcome: Number of Participants With Neurocognitive Domains Preserved at Month 9
Description: as for outcome 2
Time Frame: Month 9
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | GLIADEL
Number analyzed (Participants) | 54
Participants
  Domains preserved=3 | 14
  Domains preserved=2 | 6
  Domains preserved=1 | 0
  Domains preserved=0 | 0

6. Primary Outcome: Number of Participants With Neurocognitive Domains Preserved at Month 12
Description: Preservation of NF was defined as a decrease of less than or equal to (<=) 1 SD, any increase, or no change (0 SD) in z-score for each domain (memory domain, executive function domain, and fine motor coordination domain).
Time Frame: Month 12
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | GLIADEL
Number analyzed (Participants) | 54
Participants
  Domains preserved=3 | 9
  Domains preserved=2 | 5
  Domains preserved=1 | 0
  Domains preserved=0 | 0

7. Secondary Outcome: Percentage of Participants With Brain Tumor Recurrence (Local Recurrence, Distant Recurrence and Overall Recurrence)
Time Frame: Up to Month 12 (from baseline until evidence of neurological deterioration, had a local recurrence, withdrawn, died, lost to follow-up, or the study was closed)
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | GLIADEL
Number analyzed (Participants) | 54
percentage of participants
  Local Recurrence | 28.0
  Distant Recurrence | 48.0
  Overall Recurrence | 62.0

8. Secondary Outcome: Time to Recurrence (Local, Distant and Overall)
Time Frame: as for outcome 7
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | GLIADEL
Number analyzed (Participants) | 54
months
  Time to Local Recurrence | NA [7.5 to NA] — Median and upper limit of 95 percent (%) confidence interval were not estimable because less than 50% participants had the event.
  Time to Distant Recurrence | 8.5 [4.0 to NA] — Upper limit of 95% confidence interval was not estimable because majority of the events were censored for the analysis.
  Time to Overall Recurrence | 6.1 [3.9 to 8.5]

9. Secondary Outcome: Correlation of Tumor Recurrence With Residual Mass Effect
Time Frame: as for outcome 7
Population: PP1 population. Since only two participants had residual tumor mass, no correlation analyses were performed for recurrence and residual mass effect.
Arm/Group | GLIADEL
Number analyzed (Participants) | 0

10. Secondary Outcome: Correlation of Tumor Recurrence (Local, Distant or Overall) With NF Domain Scores
Description: The correlation between recurrence (local, distant or overall) & NF was assessed by presenting change in NF domain scores (memory domain [MD], executive function domain [EFD], fine motor coordination domain [FMCD]) after tumor recurrence (Visits X, X+1, X+2, and X+3) compared to before tumor recurrence (Visit X-1). Here 'Visit X' refers to visit at which participants had tumor recurrence, Visit X-1 refers to visit immediately before the recurrence and X+1, X+2, X+3 refers to subsequent first, second & third visit after the recurrence.NF domain z-scores were derived from participant's scores in individual neurocognitive tests using an age-adjusted &education-adjusted normative distribution of scores from an unimpaired population. Individual z-scores from related tests were averaged to determine overall z-score for each of NF domains.
Time Frame: as for outcome 7
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | GLIADEL
Number analyzed (Participants) | 54
z-score
  Local Recurrence: MD at Visit (X-1): number analyzed (Participants) | 14
  Local Recurrence: MD at Visit (X-1) | -0.9 (1.21)
  Local Recurrence: MD Change at Visit (X-1): number analyzed (Participants) | 7
  Local Recurrence: MD Change at Visit (X-1) | -1.1 (1.11)
  Local Recurrence: MD Change at Visit (X+1): number analyzed (Participants) | 4
  Local Recurrence: MD Change at Visit (X+1) | 0.7 (0.38)
  Local Recurrence: MD Change at Visit (X+2): number analyzed (Participants) | 4
  Local Recurrence: MD Change at Visit (X+2) | 0.1 (1.80)
  Local Recurrence: MD Change at Visit (X+3): number analyzed (Participants) | 1
  Local Recurrence: MD Change at Visit (X+3) | -0.8 (NA) — Standard deviation could not be calculated since only 1 participant was analyzed.
  Local Recurrence: EFD at Visit (X-1): number analyzed (Participants) | 11
  Local Recurrence: EFD at Visit (X-1) | -0.4 (1.76)
  Local Recurrence: EFD Change at Visit (X-1): number analyzed (Participants) | 6
  Local Recurrence: EFD Change at Visit (X-1) | -0.5 (0.62)
  Local Recurrence: EFD Change at Visit (X+1): number analyzed (Participants) | 4
  Local Recurrence: EFD Change at Visit (X+1) | 0.2 (0.89)
  Local Recurrence: EFD Change at Visit (X+2): number analyzed (Participants) | 4
  Local Recurrence: EFD Change at Visit (X+2) | -0.0 (0.74)
  Local Recurrence: EFD Change at Visit (X+3): number analyzed (Participants) | 1
  Local Recurrence: EFD Change at Visit (X+3) | -1.1 (NA) — Standard deviation could not be calculated since only 1 participant was analyzed.
  Local Recurrence: FMCD at Visit (X-1): number analyzed (Participants) | 14
  Local Recurrence: FMCD at Visit (X-1) | -1.5 (1.65)
  Local Recurrence: FMCD Change at Visit (X-1): number analyzed (Participants) | 8
  Local Recurrence: FMCD Change at Visit (X-1) | 0.4 (0.59)
  Local Recurrence: FMCD Change at Visit (X+1): number analyzed (Participants) | 4
  Local Recurrence: FMCD Change at Visit (X+1) | 0.5 (0.53)
  Local Recurrence: FMCD Change at Visit (X+2): number analyzed (Participants) | 4
  Local Recurrence: FMCD Change at Visit (X+2) | -0.4 (0.70)
  Local Recurrence: FMCD Change at Visit (X+3): number analyzed (Participants) | 1
  Local Recurrence: FMCD Change at Visit (X+3) | 0.3 (NA) — Standard deviation could not be calculated since only 1 participant was analyzed.
  Distant Recurrence: MD at Visit (X-1): number analyzed (Participants) | 23
  Distant Recurrence: MD at Visit (X-1) | -1.0 (1.04)
  Distant Recurrence: MD Change at Visit (X-1): number analyzed (Participants) | 19
  Distant Recurrence: MD Change at Visit (X-1) | 0.2 (1.35)
  Distant Recurrence: MD Change at Visit (X+1): number analyzed (Participants) | 11
  Distant Recurrence: MD Change at Visit (X+1) | -0.2 (1.02)
  Distant Recurrence: MD Change at Visit (X+2): number analyzed (Participants) | 5
  Distant Recurrence: MD Change at Visit (X+2) | -0.2 (1.77)
  Distant Recurrence: MD Change at Visit (X+3): number analyzed (Participants) | 2
  Distant Recurrence: MD Change at Visit (X+3) | -0.7 (0.07)
  Distant Recurrence: EFD at Visit (X-1): number analyzed (Participants) | 23
  Distant Recurrence: EFD at Visit (X-1) | -0.2 (1.44)
  Distant Recurrence: EFD Change at Visit (X-1): number analyzed (Participants) | 19
  Distant Recurrence: EFD Change at Visit (X-1) | -0.2 (0.82)
  Distant Recurrence: EFD Change at Visit (X+1): number analyzed (Participants) | 10
  Distant Recurrence: EFD Change at Visit (X+1) | -0.5 (1.11)
  Distant Recurrence: EFD Change at Visit (X+2): number analyzed (Participants) | 5
  Distant Recurrence: EFD Change at Visit (X+2) | -0.8 (1.20)
  Distant Recurrence: EFD Change at Visit (X+3): number analyzed (Participants) | 2
  Distant Recurrence: EFD Change at Visit (X+3) | -0.8 (0.39)
  Distant Recurrence: FMCD at Visit (X-1): number analyzed (Participants) | 23
  Distant Recurrence: FMCD at Visit (X-1) | -1.2 (1.32)
  Distant Recurrence: FMCD Change at Visit (X-1): number analyzed (Participants) | 18
  Distant Recurrence: FMCD Change at Visit (X-1) | -0.1 (0.61)
  Distant Recurrence: FMCD Change at Visit (X+1): number analyzed (Participants) | 10
  Distant Recurrence: FMCD Change at Visit (X+1) | -0.4 (0.99)
  Distant Recurrence: FMCD Change at Visit (X+2): number analyzed (Participants) | 5
  Distant Recurrence: FMCD Change at Visit (X+2) | -1.1 (1.03)
  Distant Recurrence: FMCD Change at Visit (X+3): number analyzed (Participants) | 2
  Distant Recurrence: FMCD Change at Visit (X+3) | -0.1 (0.48)
  Overall Recurrence: MD at Visit (X-1): number analyzed (Participants) | 30
  Overall Recurrence: MD at Visit (X-1) | -0.9 (1.15)
  Overall Recurrence: MD Change at Visit (X-1): number analyzed (Participants) | 20
  Overall Recurrence: MD Change at Visit (X-1) | -0.1 (1.40)
  Overall Recurrence: MD Change at Visit (X+1): number analyzed (Participants) | 13
  Overall Recurrence: MD Change at Visit (X+1) | -0.1 (0.96)
  Overall Recurrence: MD Change at Visit (X+2): number analyzed (Participants) | 8
  Overall Recurrence: MD Change at Visit (X+2) | -0.2 (1.67)
  Overall Recurrence: MD Change at Visit (X+3): number analyzed (Participants) | 2
  Overall Recurrence: MD Change at Visit (X+3) | -0.7 (0.07)
  Overall Recurrence: EFD at Visit (X-1): number analyzed (Participants) | 27
  Overall Recurrence: EFD at Visit (X-1) | -0.1 (1.47)
  Overall Recurrence: EFD Change at Visit (X-1): number analyzed (Participants) | 19
  Overall Recurrence: EFD Change at Visit (X-1) | -0.3 (0.76)
  Overall Recurrence: EFD Change at Visit (X+1): number analyzed (Participants) | 12
  Overall Recurrence: EFD Change at Visit (X+1) | -0.5 (1.01)
  Overall Recurrence: EFD Change at Visit (X+2): number analyzed (Participants) | 8
  Overall Recurrence: EFD Change at Visit (X+2) | -0.6 (0.98)
  Overall Recurrence: EFD Change at Visit (X+3): number analyzed (Participants) | 2
  Overall Recurrence: EFD Change at Visit (X+3) | -0.8 (0.39)
  Overall Recurrence: FMCD at Visit (X-1): number analyzed (Participants) | 30
  Overall Recurrence: FMCD at Visit (X-1) | -1.2 (1.31)
  Overall Recurrence: FMCD Change at Visit (X-1): number analyzed (Participants) | 20
  Overall Recurrence: FMCD Change at Visit (X-1) | 0.0 (0.69)
  Overall Recurrence: FMCD Change at Visit (X+1): number analyzed (Participants) | 12
  Overall Recurrence: FMCD Change at Visit (X+1) | -0.3 (0.92)
  Overall Recurrence: FMCD Change at Visit (X+2): number analyzed (Participants) | 8
  Overall Recurrence: FMCD Change at Visit (X+2) | -0.9 (0.95)
  Overall Recurrence: FMCD Change at Visit (X+3): number analyzed (Participants) | 2
  Overall Recurrence: FMCD Change at Visit (X+3) | -0.1 (0.48)

11. Secondary Outcome: Percentage of Participants With Neurologic Death
Description: Neurologic Death was defined as death due to progression of neurologic disease.
Time Frame: as for outcome 7
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | GLIADEL
Number analyzed (Participants) | 54
percentage of participants | 1.9

12. Secondary Outcome: Time to Neurocognitive Deterioration
Description: The time to neurocognitive deterioration was defined as the number of days between the date of study treatment and the date of neurocognitive deterioration based on NF assessment. This was assessed using Kaplan Meier method.
Time Frame: as for outcome 7
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: months
Arm/Group | GLIADEL
Number analyzed (Participants) | 54
months | NA [NA to NA] — Time to neurocognitive deterioration was not estimable because majority of the events were censored for the analysis.

13. Secondary Outcome: Percentage of Participants With Neurocognitive Decline in NF by Severity (Memory Domain, Executive Function Domain, and Fine Motor Coordination Domain)
Description: Neurocognitive decline was defined as any decrease in NF scores less than (<) 0 SD from baseline. Here, in category titles EFD represents Executive Function Domain and FMCD represents Fine Motor Coordination Domain.
Time Frame: Months 2, 4, 6, 9 and 12
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | GLIADEL
Number analyzed (Participants) | 54
percentage of participants
  Month 2: Memory Domain, decline <0 to -1 SD | 27.3
  Month 2: Memory Domain, decline <-1 to -2 SD | 15.9
  Month 2: Memory Domain, decline <-2 to -3 SD | 4.5
  Month 2: Memory Domain, decline <-3 to -4 SD | 0
  Month 2: Memory Domain, decline <-4 to -5 SD | 0
  Month 2: Memory Domain, decline <-5 SD | 0
  Month 2: EFD, decline <0 to -1 SD | 37.8
  Month 2: EFD, decline <-1 to -2 SD | 8.1
  Month 2: EFD, decline <-2 to -3 SD | 0
  Month 2: EFD, decline <-3 to -4 SD | 0
  Month 2: EFD, decline <-4 to -5 SD | 0
  Month 2: EFD, decline <-5 SD | 0
  Month 2: FMCD, decline <0 to -1 SD | 23.8
  Month 2: FMCD, decline <-1 to -2 SD | 7.1
  Month 2: FMCD, decline <-2 to -3 SD | 2.4
  Month 2: FMCD, decline <-3 to -4 SD | 2.4
  Month 2: FMCD, decline <-4 to -5 SD | 0
  Month 2: FMCD, decline <-5 SD | 0
  Month 4: Memory Domain, decline <0 to -1 SD | 19.4
  Month 4: Memory Domain, decline <-1 to -2 SD | 8.3
  Month 4: Memory Domain, decline <-2 to -3 SD | 0
  Month 4: Memory Domain, decline <-3 to -4 SD | 0
  Month 4: Memory Domain, decline <-4 to -5 SD | 2.8
  Month 4: Memory Domain, decline <-5 SD | 2.8
  Month 4: EFD, decline <0 to -1 SD | 29.0
  Month 4: EFD, decline <-1 to -2 SD | 0
  Month 4: EFD, decline <-2 to -3 SD | 0
  Month 4: EFD, decline <-3 to -4 SD | 0
  Month 4: EFD, decline <-4 to -5 SD | 0
  Month 4: EFD, decline <-5 SD | 0
  Month 4: FMCD, decline <0 to -1 SD | 17.1
  Month 4: FMCD, decline <-1 to -2 SD | 11.4
  Month 4: FMCD, decline <-2 to -3 SD | 0
  Month 4: FMCD, decline <-3 to -4 SD | 2.9
  Month 4: FMCD, decline <-4 to -5 SD | 0
  Month 4: FMCD, decline <-5 SD | 0
  Month 6: Memory Domain, decline <0 to -1 SD | 12.5
  Month 6: Memory Domain, decline <-1 to -2 SD | 0
  Month 6: Memory Domain, decline <-2 to -3 SD | 4.2
  Month 6: Memory Domain, decline <-3 to -4 SD | 0
  Month 6: Memory Domain, decline <-4 to -5 SD | 0
  Month 6: Memory Domain, decline <-5 SD | 0
  Month 6: EFD, decline <0 to -1 SD | 18.2
  Month 6: EFD, decline <-1 to -2 SD | 4.5
  Month 6: EFD, decline <-2 to -3 SD | 0
  Month 6: EFD, decline <-3 to -4 SD | 0
  Month 6: EFD, decline <-4 to -5 SD | 0
  Month 6: EFD, decline <-5 SD | 0
  Month 6: FMCD, decline <0 to -1 SD | 12.5
  Month 6: FMCD, decline <-1 to -2 SD | 20.8
  Month 6: FMCD, decline <-2 to -3 SD | 0
  Month 6: FMCD, decline <-3 to -4 SD | 0
  Month 6: FMCD, decline <-4 to -5 SD | 0
  Month 6: FMCD, decline <-5 SD | 0
  Month 9: Memory Domain, decline <0 to -1 SD | 25.0
  Month 9: Memory Domain, decline <-1 to -2 SD | 5.0
  Month 9: Memory Domain, decline <-2 to -3 SD | 0
  Month 9: Memory Domain, decline <-3 to -4 SD | 0
  Month 9: Memory Domain, decline <-4 to -5 SD | 0
  Month 9: Memory Domain, decline <-5 SD | 0
  Month 9: EFD, decline <0 to -1 SD | 36.8
  Month 9: EFD, decline <-1 to -2 SD | 5.3
  Month 9: EFD, decline <-2 to -3 SD | 0
  Month 9: EFD, decline <-3 to -4 SD | 0
  Month 9: EFD, decline <-4 to -5 SD | 0
  Month 9: EFD, decline <-5 SD | 0
  Month 9: FMCD, decline <0 to -1 SD | 20.0
  Month 9: FMCD, decline <-1 to -2 SD | 10.0
  Month 9: FMCD, decline <-2 to -3 SD | 5.0
  Month 9: FMCD, decline <-3 to -4 SD | 0
  Month 9: FMCD, decline <-4 to -5 SD | 0
  Month 9: FMCD, decline <-5 SD | 0
  Month 12: Memory Domain, decline <0 to -1 SD | 14.3
  Month 12: Memory Domain, decline <-1 to -2 SD | 7.1
  Month 12: Memory Domain, decline <-2 to -3 SD | 0
  Month 12: Memory Domain, decline <-3 to -4 SD | 0
  Month 12: Memory Domain, decline <-4 to -5 SD | 0
  Month 12: Memory Domain, decline <-5 SD | 0
  Month 12: EFD, decline <0 to -1 SD | 33.3
  Month 12: EFD, decline <-1 to -2 SD | 0
  Month 12: EFD, decline <-2 to -3 SD | 0
  Month 12: EFD, decline <-3 to -4 SD | 0
  Month 12: EFD, decline <-4 to -5 SD | 0
  Month 12: EFD, decline <-5 SD | 0
  Month 12: FMCD, decline <0 to -1 SD | 7.1
  Month 12: FMCD, decline <-1 to -2 SD | 14.3
  Month 12: FMCD, decline <-2 to -3 SD | 0
  Month 12: FMCD, decline <-3 to -4 SD | 0
  Month 12: FMCD, decline <-4 to -5 SD | 0
  Month 12: FMCD, decline <-5 SD | 0

ADVERSE EVENTS:
Time Frame: Screening up to 12 months
Description: The study team only has access to serious and all treatment-emergent adverse events (serious and non-serious). All efforts to locate other adverse event data have been exhausted. All treatment-emergent adverse events, whether serious or non-serious, have been reported in the Other (Not Including Serious) Adverse Events tables as severity of the event cannot be distinguished in available data.
Arm/Group | GLIADEL
All-Cause Mortality (participants affected / at risk) | 9/59
Serious Adverse Events (participants affected / at risk) | 40/59
Other Adverse Events (participants affected / at risk) | 53/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GLIADEL (N=59)
Cardiac failure congestive (Cardiac disorders) | 1
Cardiopulmonary failure (Cardiac disorders) | 1
Adrenal insufficiency (Endocrine disorders) | 1
Lip pain (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Asthenia (General disorders) | 2
Drug withdrawal syndrome (General disorders) | 1
Multi-organ failure (General disorders) | 1
Pyrexia (General disorders) | 1
Brain abscess (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 1
Device related infection (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 2
Wound infection (Infections and infestations) | 1
Haemothorax (Injury, poisoning and procedural complications) | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 1
Blood creatinine increased (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 3
Failure to thrive (Metabolism and nutrition disorders) | 6
Hyponatraemia (Metabolism and nutrition disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1
Soft tissue necrosis (Musculoskeletal and connective tissue disorders) | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 18
Metastases to adrenals (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to small intestine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neoplasm recurrence (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5
Convulsion (Nervous system disorders) | 2
Headache (Nervous system disorders) | 2
Intracranial hypotension (Nervous system disorders) | 1
Visual field defect (Nervous system disorders) | 1
Agitation (Psychiatric disorders) | 1
Anxiety (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 1
Mental status changes (Psychiatric disorders) | 1
Haematuria (Renal and urinary disorders) | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Deep vein thrombosis (Vascular disorders) | 5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GLIADEL (N=59)
Anaemia (Blood and lymphatic system disorders) | 3
Lymphadenopathy mediastinal (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Bradycardia (Cardiac disorders) | 3
Tachycardia (Cardiac disorders) | 1
Ventricular extrasystoles (Cardiac disorders) | 1
Eye pain (Eye disorders) | 1
Lacrimation increased (Eye disorders) | 1
Vision blurred (Eye disorders) | 3
Vision disturbance (Eye disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 9
Diarrhoea (Gastrointestinal disorders) | 2
Duodenal ulcer (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Faecal incontinence (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2
Hypoaesthesia oral (Gastrointestinal disorders) | 1
Loose tooth (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 9
Oral soft tissue disorder (Gastrointestinal disorders) | 1
Rectal discharge (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 4
Asthenia (General disorders) | 7
Chest pain (General disorders) | 1
Drug withdrawal syndrome (General disorders) | 1
Fatigue (General disorders) | 13
Gait disturbance (General disorders) | 1
Hunger (General disorders) | 1
Irritability (General disorders) | 1
Non-cardiac chest pain (General disorders) | 1
Oedema peripheral (General disorders) | 6
Pyrexia (General disorders) | 5
Drug hypersensitivity (Immune system disorders) | 1
Brain abscess (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 1
Candidiasis (Infections and infestations) | 3
Device related infection (Infections and infestations) | 1
Escherichia urinary tract infection (Infections and infestations) | 1
Herpes virus infection (Infections and infestations) | 1
Laryngitis (Infections and infestations) | 1
Lobar pneumonia (Infections and infestations) | 1
Oral candidiasis (Infections and infestations) | 3
Sinusitis (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 2
Wound infection (Infections and infestations) | 1
Fall (Injury, poisoning and procedural complications) | 1
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 1
Incision site complication (Injury, poisoning and procedural complications) | 1
Incision site erythema (Injury, poisoning and procedural complications) | 1
Incision site oedema (Injury, poisoning and procedural complications) | 1
Incision site pain (Injury, poisoning and procedural complications) | 2
Procedural hypertension (Injury, poisoning and procedural complications) | 1
Procedural pain (Injury, poisoning and procedural complications) | 36
Therapeutic agent toxicity (Injury, poisoning and procedural complications) | 1
Thermal burn (Injury, poisoning and procedural complications) | 1
Blood creatinine increased (Investigations) | 1
Blood glucose increased (Investigations) | 2
Blood potassium increased (Investigations) | 1
Blood pressure increased (Investigations) | 1
Breath sounds abnormal (Investigations) | 1
Cardiac murmur (Investigations) | 1
Weight decreased (Investigations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 3
Dehydration (Metabolism and nutrition disorders) | 4
Failure to thrive (Metabolism and nutrition disorders) | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 17
Hyponatraemia (Metabolism and nutrition disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 6
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2
Soft tissue necrosis (Musculoskeletal and connective tissue disorders) | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neoplasm recurrence (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Amnesia (Nervous system disorders) | 1
Aphasia (Nervous system disorders) | 4
Brain stem infarction (Nervous system disorders) | 1
Clumsiness (Nervous system disorders) | 1
Convulsion (Nervous system disorders) | 6
Coordination abnormal (Nervous system disorders) | 1
Depressed level of consciousness (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 2
Headache (Nervous system disorders) | 13
Hemianopia homonymous (Nervous system disorders) | 1
Hemiparesis (Nervous system disorders) | 2
Hypoaesthesia (Nervous system disorders) | 2
Hypokinesia (Nervous system disorders) | 1
IVth nerve paralysis (Nervous system disorders) | 1
Intracranial hypotension (Nervous system disorders) | 1
Lethargy (Nervous system disorders) | 3
Paralysis (Nervous system disorders) | 1
Peroneal nerve palsy (Nervous system disorders) | 1
Pneumocephalus (Nervous system disorders) | 1
Subdural effusion (Nervous system disorders) | 2
Agitation (Psychiatric disorders) | 2
Anxiety (Psychiatric disorders) | 4
Confusional state (Psychiatric disorders) | 3
Depression (Psychiatric disorders) | 2
Insomnia (Psychiatric disorders) | 3
Mental status changes (Psychiatric disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2
Drug eruption (Skin and subcutaneous tissue disorders) | 4
Ecchymosis (Skin and subcutaneous tissue disorders) | 1
Erythema (Skin and subcutaneous tissue disorders) | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1
Hypoaesthesia facial (Skin and subcutaneous tissue disorders) | 1
Periorbital oedema (Skin and subcutaneous tissue disorders) | 1
Petechiae (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 2
Rash pruritic (Skin and subcutaneous tissue disorders) | 1
Deep vein thrombosis (Vascular disorders) | 6
Hypertension (Vascular disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes